CLINICAL TRIAL: NCT04845893
Title: Observational Study on Treatment of Skeletal Ewing Sarcoma at Diagnosis
Brief Title: Observational Study on Skeletal Ewing's Sarcoma
Acronym: EWOss
Status: Recruiting | Type: Observational
Sponsor: Italian Sarcoma Group (Network)
Responsible Party: Sponsor
Other Study IDs: ISG-EWOss
Record Dates: First submitted 2021-04-12; First posted 2021-04-15 (Actual); Last update posted 2026-01-02 (Actual); Status verified 2025-12

CONDITIONS: Ewing Sarcoma of Bone
Keywords: Ewing Sarcoma
MeSH Terms: conditions — Sarcoma, Ewing | interventions — Surgical Procedures, Operative; Radiotherapy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Skeletal Ewing Sarcoma: This cohort include patients affected by Ewing Sarcoma of bone, referred to participating Institutions.
  Interventions: Other: Treatment of Ewings Sarcoma of bone according clinical practice (includes drugs, surgery, radiotherapy or any other received treatments)

INTERVENTIONS:
Other: Treatment of Ewings Sarcoma of bone according clinical practice (includes drugs, surgery, radiotherapy or any other received treatments) — This observational study collects all the treatments received by the patients according clinical practices or experimental trials and therefore includes drug/biological/surgical/ radiotherapy and any other applicable treatments

SUMMARY:
Observational prospective trial aimed to collect the collect demographic, clinical, surgical, pathological and molecular characteristics and treatment from patients affected by skeletal Ewing Sarcoma

DETAILED DESCRIPTION:
The Ewing sarcoma treatment is based on chemotherapy, surgery and radiotherapy. Chemotherapy, performed with a combination of several drugs, is given as primary treatment before surgery.

Surgical intervention must be performed in all cases in which it is possible to obtain an excision with free margins and with acceptable functional deficits. However, when, after surgery in case of incomplete resection, post-operative radiotherapy is used, in order to reduce the risk of local recurrence as much as possible.

Subsequently in the local treatment, a phase of maintenance chemotherapy is foreseen, the intensity of which is modulated according to the response to induction therapy.

The treatments are carried out with different programs for patients with localized disease or metastatic disease and derive from clinical trials carried out in the last 30 years.

These results are the result of national and international prospective trials which, precisely due to the rarity of the disease, took many years to execute, and it is significant to know that randomized studies were in very limited numbers, as almost all the studies were represented by studies of uncontrolled phase II Improving treatments requires the expansion of knowledge on the biological behavior of this tumor and the acquisition of as much information as possible deriving from clinical experience.

For this reason, pending the definition of a new prospective randomized trial, which will take time (approximately two years) to be made operational, it is considered useful from a scientific point of view to prospectively collect data relating to new cases of Ewing's sarcoma 'bone.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of Ewing's sarcoma of the bone
2. Diagnosis of Ewing-like sarcoma (round cell sarcoma with fusion of the EWSR1 gene with others not of the ETS family, sarcoma with CIC rearrangement or sarcoma with BCOR rearrangement)
3. Diagnosis of extraosseous Ewing's sarcoma for patients
4. Age at diagnosis <50 years
5. Assessment of the extent of the disease at onset in accordance with the European Society of Medical Oncology guidelines
6. Patients or parents oe guardians of minors who have given their written informed consent to participate in the study

Exclusion Criteria:

1. Presence of comorbid factors who can compromise the compliance of the treatment plan or the evaluation of the outcomes, including but not limited to organ pathologies that contraindicate the use of chemotherapy and psychological or social conditions that do not allow for adequate compliance treatment or adequate follow-up

Ages: 0 Years to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Patients with Ewing's sarcoma of the bone or with Ewing-like sarcoma (round cell sarcoma with fusion of the EWSR1 gene with others not of the Ewings' Tumor Sarcoma family, sarcoma with Capicua Transcriptional Repressor (CIC) rearrangement or sarcoma with BCL6 corepressor (BCOR) rearrangement
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2021-06-01 (Actual); Primary Completion 2028-05-25 (Estimated); Study Completion 2028-05-25 (Estimated)

PRIMARY OUTCOMES:
5 years Event Free Survival (EFS) | 5 years
  Onset of any event (an event is the defined as disease recurrence, death for disease or any other cause)

SECONDARY OUTCOMES:
Overall Survival (OS) | at 5 years
  Time elapsed for the diagnosis to the death for any cause
Adverse events related to the treatments in patients with age >21 years at the time of diagnosis | Every 3 weeks (Week 3, week 6, week 9, week 12, ...) up to 30 months
  Number of Participants of age >21 years with Treatment-Related Adverse Events as Assessed by CTCAE v5.0,
To assess baseline clinical and disease-specific factors with possible impact on survival analyses in the subpopulation with Ewing-like sarcoma | Baseline
  Collection of clinical pathological characteristics at disease presentation/diagnosis

CONTACTS AND LOCATIONS:
Locations (18):
- Italy (18):
  - Istituto Clinico Humanitas, Rozzano, MI
  - Centro di Riferimento Oncologico - Unit of Medical Oncology, Aviano, Pordenone
  - I.R.C.C. - Unit of Medical Oncology, Candiolo, Torino
  - Azienda ospedaliero universitaria consorziale policlinico - bari, Bari
  - A.O. Universitaria Policlinico S. Orsola Malpighi di Bologna, Bologna
  - Istituto ortopedico Rizzoli, Bologna
  - A.O. Universitaria Meyer, Florence
  - Istituto Giannina Gaslini, Genova
  - FONDAZIONE IRCCS Istituto Nazionale dei Tumori, Milan
  - Azienda Ospedaliera Santobono Pausilipon, Napoli
  - Azienda Ospedaliera di Padova, Padua
  - ARNAS P. O. "Civico e Benfratelli", Palermo
  - Azienda Ospedaliera Universitaria di Parma, Parma
  - Azienda Ospedaliero-Universitaria Pisana, Pisa
  - Ospedale Pediatrico Bambin Gesu', Roma
  - Istituto Regina Elena - IFO, Rome
  - Ospedale Infantile Regina Margherita - Unit of Paediatric Oncoematology, Torino
  - IRCCS materno infantile Burlo Garofolo, Trieste

IPD SHARING:
Plan to Share IPD: No
Not planned

REFERENCES:
- [Background] Riggi N, Suva ML, Stamenkovic I. Ewing's Sarcoma. N Engl J Med. 2021 Jan 14;384(2):154-164. doi: 10.1056/NEJMra2028910. No abstract available. PMID 33497548
- [Background] Casali PG, Bielack S, Abecassis N, Aro HT, Bauer S, Biagini R, Bonvalot S, Boukovinas I, Bovee JVMG, Brennan B, Brodowicz T, Broto JM, Brugieres L, Buonadonna A, De Alava E, Dei Tos AP, Del Muro XG, Dileo P, Dhooge C, Eriksson M, Fagioli F, Fedenko A, Ferraresi V, Ferrari A, Ferrari S, Frezza AM, Gaspar N, Gasperoni S, Gelderblom H, Gil T, Grignani G, Gronchi A, Haas RL, Hassan B, Hecker-Nolting S, Hohenberger P, Issels R, Joensuu H, Jones RL, Judson I, Jutte P, Kaal S, Kager L, Kasper B, Kopeckova K, Krakorova DA, Ladenstein R, Le Cesne A, Lugowska I, Merimsky O, Montemurro M, Morland B, Pantaleo MA, Piana R, Picci P, Piperno-Neumann S, Pousa AL, Reichardt P, Robinson MH, Rutkowski P, Safwat AA, Schoffski P, Sleijfer S, Stacchiotti S, Strauss SJ, Sundby Hall K, Unk M, Van Coevorden F, van der Graaf WTA, Whelan J, Wardelmann E, Zaikova O, Blay JY; ESMO Guidelines Committee, PaedCan and ERN EURACAN. Bone sarcomas: ESMO-PaedCan-EURACAN Clinical Practice Guidelines for diagnosis, treatment and follow-up. Ann Oncol. 2018 Oct 1;29(Suppl 4):iv79-iv95. doi: 10.1093/annonc/mdy310. No abstract available. PMID 30285218
- [Background] Gaspar N, Hawkins DS, Dirksen U, Lewis IJ, Ferrari S, Le Deley MC, Kovar H, Grimer R, Whelan J, Claude L, Delattre O, Paulussen M, Picci P, Sundby Hall K, van den Berg H, Ladenstein R, Michon J, Hjorth L, Judson I, Luksch R, Bernstein ML, Marec-Berard P, Brennan B, Craft AW, Womer RB, Juergens H, Oberlin O. Ewing Sarcoma: Current Management and Future Approaches Through Collaboration. J Clin Oncol. 2015 Sep 20;33(27):3036-46. doi: 10.1200/JCO.2014.59.5256. Epub 2015 Aug 24. PMID 26304893
- [Background] Womer RB, West DC, Krailo MD, Dickman PS, Pawel BR, Grier HE, Marcus K, Sailer S, Healey JH, Dormans JP, Weiss AR. Randomized controlled trial of interval-compressed chemotherapy for the treatment of localized Ewing sarcoma: a report from the Children's Oncology Group. J Clin Oncol. 2012 Nov 20;30(33):4148-54. doi: 10.1200/JCO.2011.41.5703. Epub 2012 Oct 22. PMID 23091096
- [Background] Ferrari S, Sundby Hall K, Luksch R, Tienghi A, Wiebe T, Fagioli F, Alvegard TA, Brach Del Prever A, Tamburini A, Alberghini M, Gandola L, Mercuri M, Capanna R, Mapelli S, Prete A, Carli M, Picci P, Barbieri E, Bacci G, Smeland S. Nonmetastatic Ewing family tumors: high-dose chemotherapy with stem cell rescue in poor responder patients. Results of the Italian Sarcoma Group/Scandinavian Sarcoma Group III protocol. Ann Oncol. 2011 May;22(5):1221-1227. doi: 10.1093/annonc/mdq573. Epub 2010 Nov 8. PMID 21059639
- [Background] Luksch R, Tienghi A, Hall KS, Fagioli F, Picci P, Barbieri E, Gandola L, Eriksson M, Ruggieri P, Daolio P, Lindholm P, Prete A, Bisogno G, Tamburini A, Grignani G, Abate ME, Podda M, Smeland S, Ferrari S. Primary metastatic Ewing's family tumors: results of the Italian Sarcoma Group and Scandinavian Sarcoma Group ISG/SSG IV Study including myeloablative chemotherapy and total-lung irradiation. Ann Oncol. 2012 Nov;23(11):2970-2976. doi: 10.1093/annonc/mds117. Epub 2012 Jul 5. PMID 22771824
- [Background] Dirksen U, Brennan B, Le Deley MC, Cozic N, van den Berg H, Bhadri V, Brichard B, Claude L, Craft A, Amler S, Gaspar N, Gelderblom H, Goldsby R, Gorlick R, Grier HE, Guinbretiere JM, Hauser P, Hjorth L, Janeway K, Juergens H, Judson I, Krailo M, Kruseova J, Kuehne T, Ladenstein R, Lervat C, Lessnick SL, Lewis I, Linassier C, Marec-Berard P, Marina N, Morland B, Pacquement H, Paulussen M, Randall RL, Ranft A, Le Teuff G, Wheatley K, Whelan J, Womer R, Oberlin O, Hawkins DS; Euro-E.W.I.N.G. 99 and Ewing 2008 Investigators. High-Dose Chemotherapy Compared With Standard Chemotherapy and Lung Radiation in Ewing Sarcoma With Pulmonary Metastases: Results of the European Ewing Tumour Working Initiative of National Groups, 99 Trial and EWING 2008. J Clin Oncol. 2019 Dec 1;37(34):3192-3202. doi: 10.1200/JCO.19.00915. Epub 2019 Sep 25. PMID 31553693
- [Background] Ladenstein R, Potschger U, Le Deley MC, Whelan J, Paulussen M, Oberlin O, van den Berg H, Dirksen U, Hjorth L, Michon J, Lewis I, Craft A, Jurgens H. Primary disseminated multifocal Ewing sarcoma: results of the Euro-EWING 99 trial. J Clin Oncol. 2010 Jul 10;28(20):3284-91. doi: 10.1200/JCO.2009.22.9864. Epub 2010 Jun 14. PMID 20547982
- [Background] Whelan J, Le Deley MC, Dirksen U, Le Teuff G, Brennan B, Gaspar N, Hawkins DS, Amler S, Bauer S, Bielack S, Blay JY, Burdach S, Castex MP, Dilloo D, Eggert A, Gelderblom H, Gentet JC, Hartmann W, Hassenpflug WA, Hjorth L, Jimenez M, Klingebiel T, Kontny U, Kruseova J, Ladenstein R, Laurence V, Lervat C, Marec-Berard P, Marreaud S, Michon J, Morland B, Paulussen M, Ranft A, Reichardt P, van den Berg H, Wheatley K, Judson I, Lewis I, Craft A, Juergens H, Oberlin O; Euro-E.W.I.N.G.99 and EWING-2008 Investigators. High-Dose Chemotherapy and Blood Autologous Stem-Cell Rescue Compared With Standard Chemotherapy in Localized High-Risk Ewing Sarcoma: Results of Euro-E.W.I.N.G.99 and Ewing-2008. J Clin Oncol. 2018 Sep 6;36(31):JCO2018782516. doi: 10.1200/JCO.2018.78.2516. Online ahead of print. PMID 30188789